CLINICAL TRIAL: NCT00555542
Title: B Cell Depletion Therapy in Rheumatoid Arthritis: An Analysis of Peripheral Blood T Cell Subsets
Brief Title: An Analysis of Peripheral Blood T Cell Subsets on Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Lai-Shan Tam, The Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RA-2006-005
Record Dates: First submitted 2007-11-07; First posted 2007-11-08 (Estimated); Last update posted 2008-05-09 (Estimated); Status verified 2008-05

CONDITIONS: Rheumatoid Arthritis
Keywords: B-cell; rituximab; Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Rituximab is administrated as 1000mg intravenous infusion on day 1 and day 15.
  Interventions: Drug: rituximab

INTERVENTIONS:
Drug: rituximab — Patients are taking stable dose of methotrexate and at least 10mg folic acid per week for at least 4 weeks. Rituximab is administrated as 1000mg intravenous infusion on day 1 and day 15. Premedication as standard prescription consists of methylprednisolone 100mg IV, Chlorpheniramine maleate(piriton 10mg IV and oral paracetamol 500mg to be given 30 minutes before each infusion of rituximab. Oral prednisolone 60mg is tob e given from day 1-6 after rituximab infusion and 30mg from day 7-13.
  Other Names: Mabthera

SUMMARY:
To study the effects of T cell in peripheral blood of patients with RA undergoing selective B cell depletion have not been studied. We analyze the B and T cell subsets in patients with active RA treated undergoing this form of treatment with rituximab.

DETAILED DESCRIPTION:
* In this open labeled prospective study, we evaluate the therapeutic efficacy and peripheral blood cellular response of rituximab in 10 patients with active RA despite conventional DMARDs therapy.
* Patients are taking stable dose of methotrexate and at least 10mg folic acid per week for at least 4 weeks. Rituximab is administrated as 1000mg intravenous infusion on day 1 and day 15. Premedication as standard prescription consists of methylprednisolone 100mg IV, Chlorpheniramine maleate(piriton 10mg IV and oral paracetamol 500mg to be given 30 minutes before each infusion of rituximab. Oral prednisolone 60mg is tob e given from day 1-6 after rituximab infusion and 30mg from day 7-13.
* In patients who relapses following the first cycle can be repeated with the second cycle must fulfill the following conditions:

  1. Patients must have responded clinically to the first infusion with improvement
  2. Other disease modifying anti-rheumatic drugs (DMARDs) are not appropriate as determined by the investigators, either they have been on them before or are ineffective or due to side effects,
  3. Patients have a disease activity score DSA>2.6
  4. At least 24 weeks since the first infusion
  5. Neutrophil count of >1.5 X 103/mcL
* The second infusion consists of rituximab 1000mg intravenous infusion on day 1 and day 15 as before and the same protocol of followed up every 4 weeks up to 52 weeks from the day of the first infusion.14 Premedication as standard prescription (consists of methylprednisolone 100mg IV, Chlorpheniramine maleate(piriton) 10mg IV and oral paracetamol 500mg to be given 30 minutes before each infusion of rituximab.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 or above
* Fulfilled the 1978 American college of Rheumatology(ACR) criteria for RA
* Seropositive for RF with RF>20 IU/ml
* Active disease despite treatment with at least 2 stable dose of DMARDs for at least 16 weeks, including MRX>10mg weekly
* 4 or more swollen and/or tender joints
* Stable dose of prednisolone<=12.5mg/day or NASID for at lease 4 weeks
* MTX>10mg/wk and folic acid>10 mg/wk for at lease 4 weeks

Exclusion Criteria:

* Little or no ability for self-care
* Used a DMARD other than MTX(Leflunomide should be wash-out with cholestyramine 4 weeks prior screening)
* Received intra-articular,intramuscular, or intravenous corticosteroids in the last 4 weeks
* Concurrent treatment with any biologics within 8 weeks
* Infected joint prosthesis during the previous 5 years
* Autoimmune disease other than RA(except concurrent Sjogren's syndrome), active rheumatoid vasculitis, and history of systemic disease associated with arthritis, chronic fatigue syndrome.
* Serious infections, such as hepatitis, pneumonia, pyelonephritis in the previous 3 months
* Any chronic infectious disease such as renal infection, chest infection with bronchiectasis or sinusitis
* Recurrent bacterial infections with encapsulated organisms, primary or secondary immunodeficiency
* Active tuberculosis requiring treatment within the previous 3 years
* Opportunistic infection such as herpes zoster within the previous 2 months
* Any evidence of active cytomegalovirus;active Pneumocystis Jirovecl;or drug-resistant atypical mycobacterial infection
* Known hypersensitivity to murine proteins
* Current signs or symptoms of severe,progressive,or uncontrolled renal,hepatic,haematological,gastrointestinal,endocrine,pulmonary,cardias,neurological,or cerebral disease
* A history of lymphoproliferative disease including lymphoma or signs suggestive of disease,such as lymphadenopathy of unusual size or location(ie,lymphadenopathy nodes,in the posterior tangle of the neck,infraclavicular epitrochlear,or periaortic areas);splenomegaly
* Any know malignant disease except basal cell carcinoma currently or in the last 5 years

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2006-07; Primary Completion 2008-05 (Actual); Study Completion 2008-05 (Actual)

PRIMARY OUTCOMES:
The proportion of patients who achieved a response according to the ACR 20 response criteria at 24 weeks and 54 weeks after the initial infusion | wk52

SECONDARY OUTCOMES:
The proportion of patients who achieved a response according to ACR50,ACR70, physician's assessment of disease activity,patient's assessment of physical function by means of a health-assessment questionnaire(HAQ),quality of life measure by SF-36 | wk52

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Kwok Ming LI, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- Department of Medicine and Therapeutics, Hong Kong, China